CLINICAL TRIAL: NCT00895492
Title: Two Year (2009-2010) Surveillance of Rotavirus Genotypes Causing Acute Diarrhea in Children Younger Than 5 Years of Age Requiring Emergency Room and Hospital Admission in Two Large Cities in Chile.
Brief Title: Two-year Surveillance of Rotavirus Genotypes Causing Acute Diarrhea in Children Younger Than 5 Years Requiring Emergency Room (ER) and Hospital Admission in Chile
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Miguel O'Ryan Gallardo, Full Professor, Microbiology and Mycology Department of Medicine Faculty, Universidad de Chile., University of Chile
Other Study IDs: Merck 2009
Record Dates: First submitted 2009-05-06; First posted 2009-05-08 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Acute Diarrheal Disease; Rotavirus Infection
Keywords: diarrhea; rotavirus; genotype; VP4; VP7
MeSH Terms: conditions — Rotavirus Infections; Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stool
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sotero del Rio: Emergency Room and Hospital based surveillance
- Van Buren: Emergency Room and Hospital based surveillance

SUMMARY:
The purpose of this study is to prospectively determine the rotavirus VP7/VP4 genotypes associated with moderate to severe disease (requiring emergency room (ER) consult or hospitalization) in a large public hospital from Valparaiso and another from Santiago.

DETAILED DESCRIPTION:
Rotavirus is the leading cause of gastroenteritis in children. Our group has developed a surveillance system for acute rotavirus diarrhea in two large hospitals in Chile since 2006. Patients visiting the ER for acute non-bloody diarrhea will be enrolled after an informed consent is signed by parents. A fresh stool sample will be collected to prospectively determine the rotavirus VP7/VP4 genotypes associated with moderate to severe disease (requiring emergency room (ER) consult or hospitalization. Stool samples will be tested for rotavirus by ELISA IDEIA - Rotavirus - OXOID. Rotavirus positive samples will be genotyped as described previously (Iturriza-Gomara et al. J. Clinical Virol 2004). Overall medical visits and hospitalizations, proportion of visits and hospitalizations caused by acute diarrhea, estimated numbers of rotavirus visits and hospitalizations will be calculated for each site. Proportion of rotavirus VP7 and VP4 genotypes will be calculated for three month periods per center. Differences in proportion will be compared by chi square and Fischer's exact test when appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Children with acute diarrhea
* Children younger than 5 years

Exclusion Criteria:

* Illiterate parents
* Chronic gastrointestinal disease

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children younger than 5 years of age with acute diarrhea or related diagnosis requiring emergency room and hospital admission in two large cities in Chile
Sampling Method: Non-Probability Sample
Enrollment: 967 (Actual)
Dates: Start 2009-05; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of rotavirus VP7 and VP4 genotypes | two years

SECONDARY OUTCOMES:
Proportion of rotavirus positive episodes | two years

CONTACTS AND LOCATIONS:
Overall Officials: Miguel L O'Ryan, MD, Principal Investigator — Microbiology and Micology Program, Faculty of Medicine, University of Chile
Locations (2):
- Chile (2):
  - Hospital Van Buren, Valparaíso, Región de Valparaíso
  - Hospital Dr Sotero del Rio, Santiago, Santiago Metropolitan

REFERENCES:
- [Background] O'Ryan M, Diaz J, Mamani N, Navarrete M, Vallebuono C. Impact of rotavirus infections on outpatient clinic visits in chile. Pediatr Infect Dis J. 2007 Jan;26(1):41-5. doi: 10.1097/01.inf.0000247104.01291.71. PMID 17195704
- [Background] O'Ryan M, Perez-Schael I, Mamani N, Pena A, Salinas B, Gonzalez G, Gonzalez F, Matson DO, Gomez J. Rotavirus-associated medical visits and hospitalizations in South America: a prospective study at three large sentinel hospitals. Pediatr Infect Dis J. 2001 Jul;20(7):685-93. doi: 10.1097/00006454-200107000-00009. PMID 11465841